CLINICAL TRIAL: NCT01548534
Title: A Phase III Randomized, Multicenter, Two Arms Double-blind Trial Versus Placebo, Evaluating the Interest of a Dietary Supplementation With Docosahexaenoic Acid (DHA) During Chemotherapy for Metastatic Breast Cancer
Brief Title: A Randomised Study of Docosahexaenoic Acid (DHA) in Metastatic Breast Cancer
Acronym: DHALYA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Judicial liquidation of the society providing dietary supplementation.
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PHRN11-PB; 2011-A01029-32 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Metastatic Breast Cancer; Progesterone Receptor Positive Tumor; Estrogen Receptor Positive Tumor; HER-2 Negative Tumor
Keywords: Metastatic Breast Cancer; First-Line chemotherapy; Taxane or Anthracycline; DHA; PUFA; Dietary supplementation; First-Line Taxane or Anthracycline based chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Dietary Supplements; Fish Oils; Plant Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHA-free arm (Placebo Comparator): Dietary supplementation with vegetable oil.
  Interventions: Dietary Supplement: Dietary supplementation with vegetable oil
- DHA arm (Experimental): Dietary supplementation with fish oil.
  Interventions: Dietary Supplement: Dietary supplementation with fish oil.

INTERVENTIONS:
Dietary Supplement: Dietary supplementation with fish oil. — Patients randomized in this arm will take 3 cans/day with fish oil : DHA is 1.56 g/d and EPA is 2.64 g/d.
  Arms: DHA arm
Dietary Supplement: Dietary supplementation with vegetable oil — Patients randomized in this arm will take 3 cans/day with vegetable oil : no DHA no EPA.
  Arms: DHA-free arm

SUMMARY:
The aim of this study is to increase, by DHA-induced chemosensitization, the activity of anticancer chemotherapy in patients with a metastatic advanced breast cancer, by a nutritional approach with marin-derived PolyUnsaturated Fatty Acids (PUFA).

DETAILED DESCRIPTION:
Local relapses and metastases make breast cancer a deadly disease. A major goal remains the improvement of treatment efficacy, meaning increasing toxicity to tumor tissue, without additional toxicity to non-tumor tissues.

The literature indicates that DHA sensitizes breast malignant tumors, but not non-tumor tissues, to chemotherapy and to radiotherapy through a variety of mechanisms. DHA enrichment of tissues can be achieved through a dietary supplementation of DHA-containing oils, such as fish oil, both in experimental animal models or in humans. Therefore, this represents an original nutritional approach to increase the activity of anticancer treatments through an enhanced specificity toward tumor tissues.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer requiring first-line taxanes or anthracyclines based chemotherapy
* HER2 negative, HR positive
* Life expectancy > 3 months
* ECOG Performance Status < or = 2 within 15 days before randomization
* Measurable and/or evaluable disease according to RECIST criteria 1.1
* Age > or = 18 years and < or = 80 years
* Body Mass Index (BMI)>17 for patients < 70 years and BMI>21 for patients > 70 years, within 15 days before randomization
* Hepatic parameters : total bilirubin strictly normal, AST and ALT < or = 3xULN (5 if liver metastases) within 15 days before randomization
* Signed written informed consent

Exclusion Criteria:

* Triple negative breast cancer or HER2 over expression
* Symptomatic central nervous system metastases
* Previous chemotherapy for metastatic breast cancer
* Obesity with BMI > 35 within 15 days before randomization
* Presence of another invasive cancer
* Uncontrolled Cardiac disease or uncontrolled hypertension
* Milk protein intolerance
* Known food allergy to fish
* Women of childbearing potential not using adequate contraceptive measures, pregnant or breast feeding.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 4 months
  PFS is defined as time from randomization to disease progression or death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | The objective response is the best objective response observed from the start of treatment to progression.
  ORR will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
Overall Survival (OS) | 3 years after last chemotherapy in study
  OS is defined as time from randomization to death due to any cause.
Time To Progression (TTP) | First progression
  TTP is defined as time from randomization to first documentation of objective tumor progression according to Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
Safety ans tolerance of dietary supplementation/chemotherapy association | 4 months
  Incidence and severity of adverse events will be assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Dietary supplementation compliance | 4 months
  Compliance will be assessed through patient's diary.
Quality Of Life (QOL) | At C1, after 4 months of chemotherapy, and at the end of chemotherapy.
  QOL will be assessed by QLQ-C30 and BR23 questionnaires.
Pain evaluation | 4 months
  Pain will be assessed by a Visual Analog Scale (VAS) and analgesic consumption.
DHA plasma level | Before dietary supplementation (at C1), and after 4 months of dietary supplementation.
  Plasma phospholipids DHA incorporation will be measured with a blood sample.
Neuropathy evaluation | 4 months
  Neuropathy will be assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bougnoux, MD, PhD, Principal Investigator — University Hospital, Tours
Locations (11):
- France (11):
  - Institut de Cancérologie de l'Ouest (ICO), Angers
  - Centre Hospitalier Jacques Coeur, Bourges
  - CHU Morvan, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier, Cholet
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Bretagne sud, Lorient
  - Clinique Guillaume de Varye, Saint-Doulchard
  - Centre Hospitalier Privé, Saint-Grégoire
  - CHU Bretonneau, Tours